CLINICAL TRIAL: NCT03530956
Title: Prospective Case Study: Adaptation Period of a Novel Motorized Ankle Prosthesis, AMPfoot 4+
Brief Title: Evaluation of a Novel Bionic Foot, AMPfoot 4+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Kevin De Pauw, Doctor of Philosophy, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SRP 17
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Prosthesis User; Cognitive Change; Physical Activity
Keywords: AMPfoot; dual-task; cognitive performance; physical performance; lower-limb prosthesis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current prosthesis (Active Comparator): A unilateral transtibial amputee will conduct experiments with the current prosthesis
  Interventions: Device: Ankle Mimicking Prosthetic Foot prototype 4+
- Novel prosthesis (Experimental): A unilateral transtibial amputee will conduct experiments with the novel prosthesis
  Interventions: Device: Ankle Mimicking Prosthetic Foot prototype 4+

INTERVENTIONS:
Device: Ankle Mimicking Prosthetic Foot prototype 4+ — The amputee will walk with AMPfoot 4+, a novel bionic foot, designed and built by an engineer of department MECH (VUB, B)

SUMMARY:
Background: Evaluating the use of a novel motorized ankle prosthesis during walking and under dual task circumstances is an important step in product development.

Objective: To iteratively evaluate the effectiveness of a novel bionic foot, the Ankle Mimicking Prosthetic device 4+ (or AMPfoot 4+), during walking.

Study design: Case study (crossover) research design.

Methods: One male subject will conduct a baseline experimental trial with the current prosthetic device and several experimental trials with the AMPfoot 4+ to evaluate the effectiveness of the novel device and investigate the adaptation period. Prior to baseline experiments, a familiarization trial will be performed to determine intra-subject variability of the dual task. An experimental trial consists of 2 walking tasks, i.e. the 6-minute walk test (6MWT) and the 10-meter walk test. The 6MWT will be combined with a cognitive task, i.e. backwards counting, to create dual task circumstances. The outcome measurements for the dual task are the distance covered and the walking speed, heart rate (HR) (Polar), rating of perceived exertion (RPE), VO2 (Cosmed K5), electro-encephalography (EEG), electro-myography (EMG), electro-cardiography (ECG), electrodermal activity (/skin conductance),accuracy and total duration of the cognitive task, BodyMedia (physical activity) and the visual analogue scale (VAS) for fatigue and comfort. A 10-meter walk test will be evaluated on duration.

Expected findings: In a first phase the novel device will probably reduce walking and cognitive performance, whereas fine-tuning the mechatronics (after several retests) should improve walking and cognitive performance during walking.

ELIGIBILITY:
Inclusion Criteria:

* unilateral transtibial (below knee) amputee
* healthy subject
* K4-level (Medicare), which means highest ambulation level

Exclusion Criteria:

* comorbidities
* pain in stump

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Walking distance of a 6 minute walk test | Through study completion, a period of 8 months
  Distance walked during a 6 minute hallway walk test
Walking speed of a 6 minute walk test | Through study completion, a period of 8 months
  Walking speed during a 6 minute walk test
Walking speed of a 10 meter walk test | Through study completion, a period of 8 months
  Walking speed during a 10 meter walk test
Duration of backward counting during walking (dual task) | Through study completion, a period of 8 months
  Duration of the cognitive task backward counting
Accuracy of backward counting during walking (dual task) | Through study completion, a period of 8 months
  Accuracy of responses of the cognitive task
Heart rate during walking tasks | Through study completion, a period of 8 months
  Heart rate during 6 minute and 10m walk tests
Rating of Perceived Exertion during walking tasks | Through study completion, a period of 8 months
  Rating of Perceived Exertion ranges from 6 (no exertion) until 20 (maximal exertion) during 6 minute and 10m walk tests. Higher values indicate a higher subjective feeling of exertion.
Oxygen consumption (VO2) during 6 minute walk test | Through study completion, a period of 8 months
  VO2 during 6 minute walk test
Visual analogue scale for fatigue during 6 min walk test | Through study completion, a period of 8 months
  Value at a scale (from 1 to 10) is provided using an X (as sign) and determines level of fatigue during walking. The higher the value the higher the level of fatigue
Visual analogue scale for comfort during 6 min walk test | Through study completion, a period of 8 months
  Value at a scale (from 1 to 10) is provided using an X (as sign) and determines level of comfort during walking. The higher the value the higher the level of comfort.
Brain activity | Through study completion, a period of 8 months
  Non-invasive electro-encephalography during walking
Muscle activity | Through study completion, a period of 8 months
  Non-invasive electro-myography during walking
Heart activity | Through study completion, a period of 8 months
  Non-invasive electro-cardiography during walking
Electrodermal activity | Through study completion, a period of 8 months
  Skin sensor during walking determines level of arousal

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No